CLINICAL TRIAL: NCT07160712
Title: Radicle Relief 24_RLN: A Randomized, Double-Blind, Placebo-Controlled Direct-to-Consumer Study Assessing the Impact of Health and Wellness Products on Pain and Related Health Outcomes.
Brief Title: Radicle Relief 24_RLN: A Study Assessing the Impact of Health and Wellness Products on Pain and Related Health Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX_P_2403_RLN
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on their assigned sex at birth and health outcome score during enrollment, then randomized to one of the study arms. Each participant will have an equal chance of being assigned to any study arm.
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' assigned study products. Participants are blinded to the study product they received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Control (Placebo Comparator): Relief Product Placebo Control
  Interventions: Dietary Supplement: Relief Product Placebo Control
- Active Product 1 (Experimental): Relief Active Product 1
  Interventions: Dietary Supplement: Relief Active Product 1
- Active Product 2 (Experimental): Relief Active Product 2
  Interventions: Dietary Supplement: Relief Active Product 2
- Active Product 3 (Experimental): Relief Active Product 3
  Interventions: Dietary Supplement: Relief Active Product 3

INTERVENTIONS:
Dietary Supplement: Relief Product Placebo Control — Participants will use their Relief Product Control as directed for a period of 6 weeks.
  Arms: Placebo Control
Dietary Supplement: Relief Active Product 1 — Participants will use their Relief Active Product 1 as directed for a period of 6 weeks.
  Arms: Active Product 1
Dietary Supplement: Relief Active Product 2 — Participants will use their Relief Active Product 2 as directed for a period of 6 weeks.
  Arms: Active Product 2
Dietary Supplement: Relief Active Product 3 — Participants will use their Relief Active Product 3 as directed for a period of 6 weeks.
  Arms: Active Product 3

SUMMARY:
A randomized, double-blind, placebo-controlled direct-to-consumer study assessing the impact of health and wellness products on pain and related health outcomes.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study conducted with adult participants, residing in the United States.

Eligible participants will (1) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome, and (2) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants for 7 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion

* Participants must meet all the following criteria:
* Adults, at least 21 years of age at the time of electronic consent, inclusive of all ethnicities, races, and gender identities
* Assigned sex at birth will determine sex-specific recruitment and surveys (male vs female) employed, when needed
* Resides in the United States
* Has the opportunity for at least 30% improvement in their primary health outcome
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion

* Individuals who report any of the following during screening will be excluded from participation:
* Report being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address and mobile phone number
* Reports current enrollment in another clinical trial
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
* Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.
* NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
* Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients.
* Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
* Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products
* Been diagnosed with Gastric Ulcerations
* Lack of reliable daily access to the internet

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2025-09-04 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Change in Pain Collective | 7 weeks
  Difference in rates of change over time in pain collective score as assessed by a collective of PROMIS Pain Interference 6A, Neuropathic Pain 5A, Nociceptive Pain 5A, and Pain Intensity 1A (scale 16-90; with higher scores corresponding to greater pain)

SECONDARY OUTCOMES:
Change in feelings of anxiety | 7 weeks
  Change in feelings of anxiety: Difference between rates of change over time as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in sleep | 7 weeks
  Change in sleep: Difference in rates of change over time in sleep score as assessed by PROMIS Sleep Disturbance 4A (scale 4-20; where higher scores correspond to higher levels of sleep disturbance)
Change in mood (emotional distress-depression) | 7 weeks
  Change in mood (emotional distress-depression): Difference in rates of change over time in emotional distress score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)

OTHER OUTCOMES:
Minimal clinically important difference (MCID) in mood (emotional distress-depression) | 7 weeks
  Minimal clinically important difference (MCID) in mood (emotional distress-depression): Likelihood of experiencing minimal clinically important difference in mood score as assessed by PROMIS Emotional Distress- Depression 4A (scale 4-20; with higher scores corresponding to greater levels of emotional distress)
Minimal clinically important difference (MCID) in sleep | 7 weeks
  Minimal clinically important difference (MCID) in sleep: Likelihood of experiencing minimal clinically important difference in sleep score as assessed by PROMIS Sleep Disturbance 4A (scale 4-20; where higher scores correspond to higher levels of sleep disturbance)
Change in Pain Intensity | 7 weeks
  Change in Pain Intensity: Difference in rates of change over time in pain intensity score as assessed by PROMIS Pain Intensity 3A (scale 0-10; with higher scores corresponding to more severe pain intensity)
Change in nociceptive pain | 7 weeks
  Change in nociceptive pain: Difference in rates of change over time in nociceptive pain score as assessed by PROMIS Nociceptive Pain 5A (scale 5-25; with higher scores corresponding to greater nociceptive pain)
Change in neuropathic pain | 7 weeks
  Change in neuropathic pain: Difference in rates of change over time in neuropathic pain score as assessed by PROMIS Neuropathic Pain 5A (scale 5-25; with higher scores corresponding to greater neuropathic pain)
Minimal clinically important difference (MCID) in feelings of anxiety | 7 weeks
  Minimal clinically important difference (MCID) in feelings of anxiety: Likelihood of experiencing minimal clinically important difference as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Minimal clinically important difference (MCID) in pain intensity | 7 weeks
  Minimal clinically important difference (MCID) in pain intensity: Likelihood of experiencing minimal clinically important difference in pain intensity, as assessed by PROMIS Pain Intensity 3A (scale 0-10; with higher scores corresponding to more severe pain intensity)
Minimal clinically important difference (MCID) in nociceptive pain | 7 weeks
  Minimal clinically important difference (MCID) in nociceptive pain: Likelihood of experiencing minimal clinically important difference in nociceptive pain as assessed by PROMIS Nociceptive Pain 5A (scale 5-25; with higher scores corresponding to greater nociceptive pain)
Minimal clinically important difference (MCID) in neuropathic pain | 7 weeks
  Minimal clinically important difference (MCID) in neuropathic pain: Likelihood of experiencing minimal clinically important difference in neuropathic pain as assessed by PROMIS Neuropathic Pain 5A (scale 5-25; with higher scores corresponding to greater neuropathic pain)
Minimal clinically important difference (MCID) in pain interference | 7 weeks
  Minimal clinically important difference (MCID) in pain interference: Likelihood of experiencing minimal clinically important difference in pain interference, as measured by PROMIS Pain interference (6-30; where lower scores indicate less pain interference).
Change in pain interference | 7 weeks
  Difference between rates of change over time, as measured by PROMIS Pain interference (6-30; where lower scores indicate less pain interference).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science
Locations (1):
- Radicle Science Inc., Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Related Info — https://www.radiclescience.com